CLINICAL TRIAL: NCT03703258
Title: Preventing Risky Drinking and PTSD After Sexual Assault: A Web-Based Intervention
Brief Title: Tools for Health and Resilience Implemented After Violence Exposure (Project THRIVE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Emily Dworkin, Acting Assistant Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005025; R00AA026317 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-10-11 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Post Traumatic Stress Disorder; Problem Drinking
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The THRIVE app involves 3 weeks of daily activities. Day 1 involves identification of activities to add to a "self-care activity list" with guidance around selecting activities that increase social contact, reduce alcohol use, and reduce avoidance. They will also complete an active-learning exercise about cognitive distortions and create a "stuck point to-do list" consisting of their cognitive distortions. In subsequent days, participants will be prompted to complete activities from both lists. They will also have access optional activities on topics such as asking for help, preventing isolation, deciding whether to disclose an assault, coping with negative reactions to disclosure, and thinking in helpful ways about social support. They will be prompted to complete brief daily surveys in the app, which will populate a symptom tracker. Participants in will have brief weekly phone contact with a coach to monitor safety and troubleshoot issues with app use.
  Interventions: Behavioral: App-based intervention
- Assessment-only control (No Intervention): The assessment-only control condition will involve access to a version of the app that includes daily surveys and a symptom tracker populated by these surveys, but without any of the other exercises included in the experimental version of the app. Participants in the control condition will have brief weekly phone contact with a coach to monitor safety and troubleshoot issues with app use.

INTERVENTIONS:
Behavioral: App-based intervention — A app-based cognitive-behavioral intervention to prevent the development of PTSD and high-risk drinking in recently-victimized adults
  Other Names: THRIVE app
  Arms: Intervention

SUMMARY:
Sexual assault victimization is a common and particularly harmful form of trauma that is associated with increased risk for high-risk drinking and other conditions of public health concern, such as PTSD. Given evidence that sexual assault survivors who have low social support or receive negative social reactions to sexual assault disclosure are more likely to experience PTSD and drinking problems, improving social support is a novel target for intervention. The proposed study will attempt to prevent the onset of high-risk drinking and PTSD in sexual assault survivors by developing and testing a web-based early intervention aimed at increasing contact with social supporters and mitigating the harm of negative social reactions; ultimately, results will contribute to advancing the field's understanding of the potential for social support to mitigate the harm of trauma.

DETAILED DESCRIPTION:
This study involves developing, modifying, and preliminarily testing an intervention to prevent high-risk drinking and PTSD in women who have experienced sexual assault (SA) in the past 10 weeks. In the pilot trial phase of this study, intervention feasibility will be tested in an open trial with N = 40 women with past-10-week SA histories, active drinking, and elevated distress. Participants will complete surveys at baseline, termination, and 3-month follow-up. Participants will be randomized to either the intervention (N = 20) or assessment-only control (N = 20). We hypothesize that (H1) most participants will respond positively on items assessing satisfaction with the intervention, (H2) participants will report above-average usability on a standardized measure, (H3) completion rates for daily activities will be similar to previous web-based interventions, (H4) participants will show significant learning as evidenced by increases in correct responses to knowledge questions from baseline to post, and (H5) participants in the intervention condition will evidence less high-risk drinking and PTSD at 3-month follow-up than participants in the assessment-only condition.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* self-identification as female
* sexual assault, defined as endorsement of unwanted, attempted or completed sexual contact in the past 10 weeks
* age > 18
* English fluency
* smartphone and internet access at least daily for 3 weeks and at least weekly for 3 months
* consumption of >1 alcoholic drink in the past month
* >1 episode of high-risk drinking in past 6 months, defined as either more than 3 drinks on a given day or more than 7 drinks in a given week
* at least 3 symptom clusters endorsed on the PTSD Checklist.

Exclusion Criteria:

* active suicidality
* psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who self-identify as female are eligible to participate.
Enrollment: 41 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dworkin, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Medicine, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howe ES, Dworkin ER. The day-to-day relationship between posttraumatic stress symptoms and social support after sexual assault. Eur J Psychotraumatol. 2024;15(1):2311478. doi: 10.1080/20008066.2024.2311478. Epub 2024 Feb 20. PMID 38376992
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783
- [Derived] Dworkin ER, Schallert M, Lee CM, Kaysen D. mHealth Early Intervention to Reduce Posttraumatic Stress and Alcohol Use After Sexual Assault (THRIVE): Feasibility and Acceptability Results From a Pilot Trial. JMIR Form Res. 2023 Jul 4;7:e44400. doi: 10.2196/44400. PMID 37402144
- [Derived] Dworkin ER, Schallert M, Lee CM, Kaysen D. Pilot randomized clinical trial of an app-based early intervention to reduce PTSD and alcohol use following sexual assault. Psychol Trauma. 2024 Dec;16(Suppl 3):S668-S678. doi: 10.1037/tra0001460. Epub 2023 Apr 3. PMID 37011153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January 13th, 2021 to August 24th, 2021 via mass emails sent to registered students at the University of Washington, flyers, social media ads, and provider referrals.
Pre-assignment Details: Participants were considered to be enrolled in the study once they provided informed consent at baseline. They completed the baseline assessment to confirm eligibility. Participants found to be eligible at baseline were automatically randomized.
Groups:
- Intervention: Participants in the intervention condition completed 3 weeks of daily activities and symptom self-monitoring in the THRIVE app. Day 1 involved identification of activities to add to a "self-care activity list" with guidance around selecting activities that increase social contact, reduce alcohol use, and reduce avoidance. They also completed an active-learning exercise about cognitive distortions and created a "stuck point to-do list" consisting of their cognitive distortions. In subsequent days, participants were prompted to complete activities from both lists. They also had access to optional activities on topics such as asking for help, preventing isolation, deciding whether to disclose an assault, coping with negative reactions to disclosure, and thinking in helpful ways about social support. They were prompted to complete brief daily surveys in the app, which populated a symptom tracker. Participants had brief weekly phone contact with a coach to monitor safety and troubleshoot issues with app use.
- Assessment-only Control: Participants in the control condition completed 3 weeks symptom self-monitoring. They had access to a version of the app that included daily surveys and a symptom tracker populated by these surveys, but without any of the other exercises included in the experimental version of the app. Participants had brief weekly phone contact with a coach to monitor safety and troubleshoot issues with app use.
Period: Overall Study
Arm/Group | Intervention | Assessment-only Control
Started | 20 | 21
Completed | 20 (Completed at least one of two follow-up assessments) | 21 (Completed at least one of two follow-up assessments)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Assessment-only Control | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.45 (4.31) | 20.14 (2.15) | 20.78 (3.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 12 | 6 | 18
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Problem Drinking Scores at Baseline and 3 Weeks
Description: Sum scores on Rutgers Alcohol Problem Index- Short Form (RAPI-S), which assesses alcohol use consequences. Range: 0-64; higher scores indicate worse outcome.
Time Frame: Baseline, post-intervention (3 weeks after baseline)
Population: Missing data are present at post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 12.40 (8.40) | 11.00 (6.43)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 10.16 (10.00) | 7.62 (6.26)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; p = .60, Mixed Models Analysis; Slope = 0.14, Standard Error of Mean 0.26 — Condition x time interaction coefficient from mixed-effect model using negative binomial distribution. Intervention = 1 and control = 0
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; Cohen's D = 0.36 — Between-group Cohen's d; calculated as within-group d(intervention) - within group d(control). Standardized using the standard deviation of the change scores. Negative values favor intervention and positive values favor control

2. Primary Outcome: Problem Drinking Scores at Baseline and 3 Months
Description: as for outcome 1
Time Frame: Baseline, 3 month follow-up
Population: Missing data are present at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 12.40 (8.40) | 11.00 (6.43)
  3 months: number analyzed (Participants) | 20 | 20
  3 months | 5.75 (4.69) | 5.55 (5.88)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; p = .94, Mixed Models Analysis; Slope = -0.02, Standard Error of Mean 0.27 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; Cohen's D = -0.01 — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Posttraumatic Stress Symptom Severity Score at Baseline and 3 Weeks
Description: Sum scores on the Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders-5 (PCL-5), which assesses posttraumatic stress symptom severity. Range: 0-80; higher scores indicate worse outcome.
Time Frame: Baseline, post-intervention (3 weeks after baseline)
Population: Missing data are present at post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 46.60 (11.45) | 39.81 (12.22)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 36.53 (14.00) | 35.62 (15.96)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; p = .38, Mixed Models Analysis; Slope = -0.12, Standard Error of Mean 0.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; Cohen's D = -0.15 — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Posttraumatic Stress Symptom Severity Score at Baseline and 3 Months
Description: as for outcome 3
Time Frame: Baseline, 3 month follow-up
Population: Missing data are present at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 46.60 (11.45) | 39.81 (12.22)
  3 months: number analyzed (Participants) | 20 | 20
  3 months | 22.10 (11.56) | 25.30 (15.81)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; p = .04, Mixed Models Analysis; Slope = -0.28, Standard Error of Mean 0.14 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Test type: Superiority; Cohen's D = -0.70 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Anxiety
Description: Sum scores on Generalized Anxiety Disorder-7 (GAD-7), which assesses symptoms of anxiety. Range: 0-21; higher scores indicate worse outcome.
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 13.35 (4.52) | 12.14 (5.34)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 11.32 (5.69) | 11.33 (6.49)
  3 months: number analyzed (Participants) | 19 | 20
  3 months | 9.05 (6.71) | 8.80 (5.48)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .51, Mixed Models Analysis; Slope = -1.23, Standard Error of Mean 1.88 — Post-intervention condition x time interaction coefficient from mixed-effect model using negative binomial distribution. Intervention = 1 and control = 0
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .64, Mixed Models Analysis; Slope = -0.90, Standard Error of Mean 1.90 — 3 month condition x time interaction coefficient from mixed-effect model using negative binomial distribution. Intervention = 1 and control = 0
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = -0.10 — Post-intervention between-group Cohen's d; calculated as within-group d(intervention) - within group d(control). Standardized using the standard deviation of the change scores. Negative values favor intervention and positive values favor control
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = 0.02 — 3 month between-group Cohen's d; calculated as within-group d(intervention) - within group d(control). Standardized using the standard deviation of the change scores. Negative values favor intervention and positive values favor control

6. Secondary Outcome: Coping Self-efficacy
Description: Mean scores on the Trauma Coping Self-Efficacy Scale (CSE-T), which assesses one's perceived ability to manage the demands of recovering from a potentially-traumatic event. Range: 1 to 7; higher scores indicate better outcome.
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 3.59 (0.63) | 4.00 (0.76)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 4.31 (0.79) | 4.15 (1.05)
  3 months: number analyzed (Participants) | 19 | 20
  3 months | 4.96 (1.00) | 5.08 (1.31)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .04, Mixed Models Analysis; Slope = 0.64, Standard Error of Mean 0.30 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .34, Mixed Models Analysis; Slope = 0.29, Standard Error of Mean 0.30 — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = 0.92 — Post-intervention between-group Cohen's d; calculated as within-group d(intervention) - within group d(control). Standardized using the standard deviation of the change scores. Positive values favor intervention and negative values favor control
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = 0.68 — 3 month between-group Cohen's d; calculated as within-group d(intervention) - within group d(control). Standardized using the standard deviation of the change scores. Positive values favor intervention and negative values favor control

7. Secondary Outcome: Depression
Description: Sum scores on the Patient Health Questionnaire-8 (PHQ-8), which assesses symptoms of depression. Range: 0-24; higher scores indicate worse outcome.
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 14.30 (5.73) | 10.81 (5.14)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 11.26 (6.69) | 10.14 (5.58)
  3 months: number analyzed (Participants) | 19 | 20
  3 months | 9.16 (6.72) | 7.65 (6.06)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .13, Mixed Models Analysis; Slope = -2.46, Standard Error of Mean 1.63 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .24, Mixed Models Analysis; Slope = -1.94, Standard Error of Mean 1.64 — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = -0.41 — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = -0.23 — [estimate comment as in outcome 5, analysis 4]

8. Secondary Outcome: Alcohol Consumption (Quantity)
Description: Number of drinks per week reported on the Daily Drinking Questionnaire
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
drinks per week
  Baseline | 9.35 (7.38) | 11.10 (6.79)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 7.68 (7.81) | 9.57 (6.79)
  3 months: number analyzed (Participants) | 20 | 20
  3 months | 6.25 (5.50) | 7.70 (5.90)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .85, Mixed Models Analysis; Slope = -0.05, Standard Error of Mean 0.25 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .96, Mixed Models Analysis; Slope = 0.01, Standard Error of Mean 0.25 — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = -0.15 — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = 0.003 — [estimate comment as in outcome 5, analysis 4]

9. Secondary Outcome: Alcohol Consumption (Frequency)
Description: Number of drinking days per week reported on the Daily Drinking Questionnaire
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: drinking days per week
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
drinking days per week
  Baseline | 2.90 (1.83) | 2.76 (1.48)
  Post-intervention | 2.37 (1.61) | 2.47 (1.36)
  3 months | 2.30 (1.81) | 2.35 (1.81)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .75, Mixed Models Analysis; Slope = -0.08, Standard Error of Mean 0.26 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .64, Mixed Models Analysis; Slope = -0.12, Standard Error of Mean 0.27 — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = -0.12 — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = -0.16 — [estimate comment as in outcome 5, analysis 4]

10. Secondary Outcome: Alcohol Consumption (Hours)
Description: Hours spent drinking per week reported on the Daily Drinking Questionnaire
Time Frame: Baseline, post-intervention (3 weeks after baseline), 3 month follow-up
Population: Missing data are present at post-intervention and 3 months
Measure: Mean (Standard Deviation); unit: drinking hours per week
Arm/Group | Intervention | Assessment-only Control
Number analyzed (Participants) | 20 | 21
drinking hours per week
  Baseline | 8.15 (8.03) | 8.33 (5.76)
  Post-intervention: number analyzed (Participants) | 19 | 21
  Post-intervention | 6.84 (7.13) | 7.14 (6.62)
  3 months: number analyzed (Participants) | 20 | 20
  3 months | 5.75 (5.24) | 10.15 (16.26)
Statistical Analysis 1: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; p = .86, Mixed Models Analysis; Slope = 0.06, Standard Error of Mean 0.35 — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; p = .55, Mixed Models Analysis; Slope = -0.22, Standard Error of Mean 0.36 — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Intervention vs Assessment-only Control; Baseline to post-intervention only; Test type: Superiority; Cohen's D = -0.04 — [estimate comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: Intervention vs Assessment-only Control; Baseline to 3 months; Test type: Superiority; Cohen's D = -0.39 — [estimate comment as in outcome 5, analysis 4]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention | Assessment-only Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03703258/Prot_SAP_ICF_000.pdf